CLINICAL TRIAL: NCT06995729
Title: A PHASE 1, MULTICENTER, OPEN-LABEL, SINGLE-DOSE STUDY TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF ZAVEGEPANT IN CHILDREN 6 TO LESS THAN 12 YEARS OF AGE WITH HISTORY OF MIGRAINE
Brief Title: A Study to Learn About the Study Medicine Called Zavegepant (PF-07930207) in Children With a History of Migraine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C5301023
Record Dates: First submitted 2025-05-07; First posted 2025-05-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Treatment of Migraine
Keywords: migraine; zavegepant; pediatric
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zavegepant (Experimental): Experimental medicine under study
  Interventions: Drug: Zavegepant

INTERVENTIONS:
Drug: Zavegepant — Zavegepant 5 mg or 10 mg (dose is weight-dependent)

SUMMARY:
The purpose of the study is to learn about safety and how the body processes the study medicine called Zavegepant (PF-07930207) in children with a history of migraine. This study helps understand how the medicine is changed and removed from the body after taking it.

This study is seeking participants who:

* Are children aged between 6 and less than 12 years old
* Have had migraine for at least 6 months.
* Weigh more than 15 kilograms

All participants in this study will receive zavegepant as a nasal spray once (one spray into one nostril). The dose of the study medicine that each participant receives will depend on how much the participant weighs.

The study will look at the experiences of the participants receiving the study medicine and collect data to better understand the possible benefits and unwanted effects of different doses of the study medicine.

Participants will take part in this study for up to 10 weeks. During this time, they will have 3 study visits at the study clinic, and 2 follow-up phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 6 years to less than 12 years.
2. Documented medical history of migraine with or without aura for at least 6 months before the Screening Visit.
3. Weight >15 kg at the Screening Visit

Exclusion Criteria:

1. Evidence or history of clinically significant disease.
2. Continuous migraine (defined as an unrelenting headache) within 1 month prior to Screening Visit.
3. Atypical migraine types, complications of a migraine, or a confounding and clinically significant pain syndrome.
4. Conditions that may affect the administration or absorption of the nasal product
5. Any psychiatric condition that is uncontrolled and/or untreated, including:

   * Clinically significant depression (Promis Parent Proxy SF 2.0 Depressive Scale T score ≥70)
   * Suicidal ideation and behaviour (C-SSRS: any "yes" to items 2 to 5 or any "yes" to suicide behaviours)
6. Serum Total bilirubin >1.5 × ULN (Upper Limit of Normal), AST (Aspartate Transferase) or ALT (Alanine Transaminase) >2 × ULN
7. Abnormal ECG (Electrocardiogram) at screening visit

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-08-12 (Estimated); Study Completion 2027-08-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1: 0 hour, 1.25 hours, 3.5 hours; Day 2: 18 hours
  Cmax is defined as the maximum observed plasma concentration of zavegepant after administration of a single dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1: 0 hour, 1.25 hours, 3.5 hours; Day 2: 18 hours
  Tmax is defined as the time to reach maximum observed plasma concentration
Area Under the Curve From Time Zero to infinity. | Day 1: 0 hour, 1.25 hours, 3.5 hours; Day 2: 18 hours
  AUC (0 - inf) is defined as area under the concentration-time curve from time 0 to infinity.

SECONDARY OUTCOMES:
Number of Participants with All-Causality Treatment-emergent Adverse Events (TEAEs) | TEAE is reported from informed consent up to 28 days after administration of study drug.
  An AE is any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship with the study intervention. SAE is defined as one of the following: is fatal or life threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Number of participants with clinically significant abnormal vital signs | Assessed from screening up to 6 days after administration of study drug
  Vital sign measurements include temperature, respiratory rate, pulse rate, and blood pressure.
Number of participants with clinically significant abnormal laboratory findings | Assessed from screening up to 6 days after administration of study drug
  Laboratory assessment includes hematology, chemistry and urinalysis. Clinical significance of laboratory abnormalities was judged by investigator.
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | Assessed from screening up to 6 days after administration of study drug
  The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. The C-SSRS assessment MUST be performed by an adequately trained, certified, and delegated rater. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts toward imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), 4: any suicidal behavior or ideation, suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior").

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Velocity Clinical Research, Washington DC, Washington D.C., District of Columbia
  - Coastal Heritage Clinical Research, Hinesville, Georgia
  - Clinical Research Institute, Minneapolis, Minnesota
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - True North Neurology, Port Jefferson Station, New York
  - Accellacare - Piedmont, Statesville, North Carolina
  - Accellacare of Piedmont HealthCare, Statesville, North Carolina
  - Central States Research, Tulsa, Oklahoma
  - Cedar Health Research, Dallas, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Granger Medical Holladay - Holladay Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301023